CLINICAL TRIAL: NCT01861808
Title: Investigation on the Prognostic Value of Biochemical Markers in the Cerebrospinal Fluid for the Functional Outcome of Spinal Cord Injured Patients
Brief Title: Prognostic Value of Biochemical Markers in Cerebrospinal Fluid for Functional Outcome of Spinal Cord Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CE 12105; RF-2010-2315118 (Other: Identification number assigned by Ethics Committee)
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Cerebrospinal Fluid
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lumbar puncture (Other): That's not really an arm label because the only intervention on the patients is the lumbar puncture
  Interventions: Other: Lumbar puncture

INTERVENTIONS:
Other: Lumbar puncture — The only intervention is the lumbar puncture on the patients to obtain a Cerebrospinal Fluid sample

SUMMARY:
The project is aimed to develop predictive indices of spinal cord injury severity through the analysis of cerebrospinal fluid of patient collected during acute injury.

ELIGIBILITY:
Inclusion Criteria:

* presence of cervical and thoracic Spinal Cord Injury
* need to be submitted to spine surgical stabilization with posterior approach

Exclusion Criteria:

* prior to recruitment, in the acute phase, treatment with steroid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08-24 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Creation of a model which analyze relationship among laboratory investigations and primary lesion, secondary damage and functional impairment | Three years
  Correlation of the dosage of more than 20 tentative biomarkers with the biological effect of Cerebrospinal Fluid exposure on human cell lines, in order to directly test those effects.
  The Cerebrospinal Fluid will be encoded using technical procedures, divided into aliquots, quickly frozen and stored at 80°C.
  Biomarkers will be measured in the Cerebrospinal Fluid, related to:
  * inflammatory and vascular reaction, by a cytokine panel including 12 different cytokines/chemochines;
  * neurodegeneration and excitotoxicity, by a panel of 10 different biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Gordini, MD, Principal Investigator — Azienda Unità Sanitaria Locale Bologna
Locations (4):
- Italy (4):
  - Montecatone Rehabilitation Institute SpA, Imola, Bologna
  - Centro Interdipartimentale Ricerca Industriale Università degli Studi, Ozzano Monferrato, Bologna
  - UOC Rianimazione CO e 118 Ospedale Maggiore AUSL, Bologna
  - UOSD Chirurgia Vertebrale di Urgenza e del Trauma Ospedale Maggiore AUSL, Bologna

REFERENCES:
- [Background] Dumont RJ, Verma S, Okonkwo DO, Hurlbert RJ, Boulos PT, Ellegala DB, Dumont AS. Acute spinal cord injury, part II: contemporary pharmacotherapy. Clin Neuropharmacol. 2001 Sep-Oct;24(5):265-79. doi: 10.1097/00002826-200109000-00003. PMID 11586111
- [Background] Lubieniecka JM, Streijger F, Lee JH, Stoynov N, Liu J, Mottus R, Pfeifer T, Kwon BK, Coorssen JR, Foster LJ, Grigliatti TA, Tetzlaff W. Biomarkers for severity of spinal cord injury in the cerebrospinal fluid of rats. PLoS One. 2011 Apr 29;6(4):e19247. doi: 10.1371/journal.pone.0019247. PMID 21559420
- [Background] Kwon BK, Stammers AM, Belanger LM, Bernardo A, Chan D, Bishop CM, Slobogean GP, Zhang H, Umedaly H, Giffin M, Street J, Boyd MC, Paquette SJ, Fisher CG, Dvorak MF. Cerebrospinal fluid inflammatory cytokines and biomarkers of injury severity in acute human spinal cord injury. J Neurotrauma. 2010 Apr;27(4):669-82. doi: 10.1089/neu.2009.1080. PMID 20038240
- [Background] Kwon BK, Casha S, Hurlbert RJ, Yong VW. Inflammatory and structural biomarkers in acute traumatic spinal cord injury. Clin Chem Lab Med. 2011 Mar;49(3):425-33. doi: 10.1515/CCLM.2011.068. Epub 2010 Dec 23. PMID 21175377
- [Background] Oyinbo CA. Secondary injury mechanisms in traumatic spinal cord injury: a nugget of this multiply cascade. Acta Neurobiol Exp (Wars). 2011;71(2):281-99. doi: 10.55782/ane-2011-1848. PMID 21731081
- [Background] Pajoohesh-Ganji A, Byrnes KR. Novel neuroinflammatory targets in the chronically injured spinal cord. Neurotherapeutics. 2011 Apr;8(2):195-205. doi: 10.1007/s13311-011-0036-2. PMID 21394541
- [Background] Rossignol S, Schwab M, Schwartz M, Fehlings MG. Spinal cord injury: time to move? J Neurosci. 2007 Oct 31;27(44):11782-92. doi: 10.1523/JNEUROSCI.3444-07.2007. PMID 17978014
- [Background] Sekhon LH, Fehlings MG. Epidemiology, demographics, and pathophysiology of acute spinal cord injury. Spine (Phila Pa 1976). 2001 Dec 15;26(24 Suppl):S2-12. doi: 10.1097/00007632-200112151-00002. PMID 11805601
- [Background] Tsai MC, Wei CP, Lee DY, Tseng YT, Tsai MD, Shih YL, Lee YH, Chang SF, Leu SJ. Inflammatory mediators of cerebrospinal fluid from patients with spinal cord injury. Surg Neurol. 2008 Dec;70 Suppl 1:S1:19-24; discussion S1:24. doi: 10.1016/j.surneu.2007.09.033. PMID 19061765
- [Background] van den Berg ME, Castellote JM, Mahillo-Fernandez I, de Pedro-Cuesta J. Incidence of spinal cord injury worldwide: a systematic review. Neuroepidemiology. 2010;34(3):184-92; discussion 192. doi: 10.1159/000279335. Epub 2010 Feb 2. PMID 20130419